CLINICAL TRIAL: NCT03701451
Title: Clinical Efficacy Observation of Demethylated Drug Decitabine in the Treatment of Locally Advanced Nasopharyngeal Carcinoma
Brief Title: Demethylated Drug in the Treatment of Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wei Jiang (Other)
Collaborators: Guilin Hospital of Traditional Chinese Medicine (Unknown)
Responsible Party: Sponsor-Investigator, Wei Jiang, Wei Jiang, MD, PhD, Guilin Medical University, China
Organization: Guilin Medical University, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLMU-05
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; Decitabine; Concurrent chemoradiotherapy; Induced chemotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- decitabin and cisplatin induced chemotherapy followed by CC (Experimental): Treated by demethylated drug decitabine injection combined with cisplatin induced chemotherapy followed by concurrent chemoradiotherapy
  Interventions: Drug: Demethylated drug decitabine

INTERVENTIONS:
Drug: Demethylated drug decitabine — Induced treatment by demethylating drug decitabine 7mg/m2 d1-5 and cisplatin 80mg/m2 d1 for 3 cycles to regionally advanced nasopharyngeal carcinoma followed by concurrent chemoradiotherapy with cisplatin 80mg/m2 d1 for 3 cycles.

SUMMARY:
The study is to observe the efficacy and toxicity of demethylating drug decitabine and cisplatin induced chemotherapy for 3 cycles followed by concurrent chemoradiotherapy in the treatment of regionally advanced nasopharyngeal carcinoma,followed up for 2 years, observing the 2-year survival rate and variation of degrees of methylation before and after treatment,providing clinical basis for the clinical study of stage II-III.

DETAILED DESCRIPTION:
Recent studies and previous studies in the investigator's research group have found that nasopharyngeal carcinoma is a disease with hypermethylation changes, and epigenetic treatment has not yet been carried out in nasopharyngeal carcinoma. In this study, Simon's two-stage design method was used to select 30 patients with nasopharyngeal carcinoma, treated with demethylating drug decitabine 7mg/m2 d1-5 + cisplatin 80mg/m2 d1 induced chemotherapy for 3 cycles followed by concurrent chemoradiotherapy with cisplatin 80mg/m2. observing the efficacy and toxicity of decitabine in the treatment of regionally advanced nasopharyngeal carcinoma, followed up for 2 years, observing the 2-year survival rate,evluating the relationship between different degrees of methylation and survival before and after treatment,provide clinical basis for the clinical study of stage II-III.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly confirmed non-keratinized or undifferentiated carcinoma of the nasopharynx.
2. Aequate hematological function: WBC ≥ 4 × 10^9 / L before the enrollment, PLT ≥ 100 × 10^9 / L, HGB ≥ 80.0g / L.
3. Adequete liver function:(serum transminase ≤ 2.5 times higher than upper limit ), renal function:(creatinine clearance rate ≥ 60 ml / min).
4. Karnofsky performance status(KPS) score of at least 70 or Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Patients must give signed infomed consent.

Exclusion Criteria:

1. Other or mixed pathological type.
2. age >65years.
3. severe heart,liver,and kidney damage.
4. histology of other malignancy .
5. prior chemotherapy or radiation of the primary tumor;Pregnant or lactating women.
6. History of psychiatric disorders .
7. Positive urine protein.
8. A healed wound for long time or incomplete fracture.
9. Before treatment,MRI showed that the tumor might be an important risk factor (for example, wrapping around the internal carotid artery / vein); or researchers judged that the tumor is a high risk of serious blood vessel bleeding during the treatment.
10. Patient who has high blood pressure can not be controlled by a single antihypertensive drug treatment (Systolic pressure > 140 mmHg, diastolic pressure > 90 mmHg.
11. Any unstable angina pectoris;with a history of angina pectoris were newly diagnosed with angina pectoris within 3 months before screening; any myocardial infarction events occurred within 6 months before screening; arrhythmia (including QTcF: male ≥ 450ms, female ≥ 470 ms) need long time use of antiarrhythmic drugs and heart function insufficiency ≥II according to New York Heart Association class.
12. Medical history of arteriovenous thrombosis event within the past year, such as cerebral vascular accident (including transient ischemic attack) and deep venous thrombosis (venous catheter thrombosis caused by chemotherapy and investigator judged that the patient had recovered, these patients should be except) and pulmonary embolism.
13. Patient who has serious hemorrhages, any serious bleeding events classification at 3 degree or more (according to CTCAE4.0) within the last 4 weeks.
14. Patient who has abnormal coagulation and bleeding tendency (signed informed consent before 14 days, and must be satisfied: INR is in the normal range without the use of anticoagulants); Application of anticoagulants or vitamin K antagonists such as Hua Falin, heparin or its analogues, with international normalized ratio (INR) is less than 1.5, allows the use of small dose Hua Falin (1 mg orally, once daily) or small dose aspirin (total dose ≤ 100 mg daily).
15. For females:patients should be surgical sterilization or postmenopausal patients, or willing to receive a medical approved contraception during treatment and 6 months after the end of the treatment; serum or urine pregnancy test must be negative, and must be non lactating period within 7 days before study; for males: patients should be treated with surgical sterilization or willing to receive a medical approved contraception during treatment and 6 months after the end of the treatment.
16. Any factors that affect the oral drug, such as the inability to swallow, diarrhea and intestinal obstruction.
17. Medical history of immunodeficiency, or other acquired, congenital immunodeficiency disease, or history of organ transplantation.
18. Any serious harm to the subject's safety or evidence of significant medical illness that in the investigator's judgment will substantially increase the risk associated with the subject's participation in and completion of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-02-28 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2 years
  The time from the first day of therapy to death or last follow-up

SECONDARY OUTCOMES:
Overall survival | 2 years
  The time from the first day of therapy to death or last follow-up
Locoregional recurrence-free survival | 2 years
  The time from the first day of therapy to death or last follow-up
Distant metastasis-free survival | 2 years
  The time from the first day of therapy to death or last follow-up
Dgree of methylation Carcinoma | 2 months
  The variations of the dgree of methylation before and after 2 months treatment
Treatment toxicity | 2moths to 2 years
  The time from the first day of therapy to death or last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Wei Jiang, PhD, Study Director — Guilin Medical University, China
Locations (2):
- China (2):
  - Guilin Hospital of Traditional Chinese Medicine, Guilin, Guangxi
  - Guilin Medical University, Guilin, Guangxi